CLINICAL TRIAL: NCT02324868
Title: Comparison of Showerpatch Versus Other Measures to Protect Intravenous Catheter Entry Site During Bathing Activities
Brief Title: Impact of Availability of Showerpatch for Patients With Intravenous Catheters
Acronym: ISIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: logistic problems
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: BEDAL (Unknown); Remedus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: S57372; FC13145773 (Other Grant/Funding Number: Flander's care)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-01

CONDITIONS: Cystic Fibrosis; Pulmonary Hypertension; Neoplasms
Keywords: Bandages; Catheter
MeSH Terms: conditions — Cystic Fibrosis; Hypertension, Pulmonary; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shower patch IV catheter protection (Experimental): Newly developed waterproof catheter dressing may be used for bathing activities
  Interventions: Device: Shower patch IV catheter protection
- Conventional IV catheter protection (Other): No specific dressing will be provided to the patient to protect the catheter entry site during bathing activities.
  Interventions: Device: Conventional IV catheter protection

INTERVENTIONS:
Device: Shower patch IV catheter protection — Shower patch will be available for the patient for bathing activities
  Arms: Shower patch IV catheter protection
Device: Conventional IV catheter protection — No Shower patch will be provided during study period
  Arms: Conventional IV catheter protection

SUMMARY:
Venous catheters are necessary for the treatment of many patients. Showering with a venous catheter is often prohibited due to the infection risk when the insertion site becomes wet. Therefore these patients are challenged to keep the catheter insertion site dry and always covered with a dressing. Washing themselves is often impossible without assistance of a nurse or significant other. For patients with a catheter connected to an infusion line, it is even more difficult. Showerpatch is a newly developed dressing that safeguards the insertion site of an IV catheter from water during bathing activities. The purpose of this trial is to evaluate the impact of the availability of Showerpatch by comparing the outcomes in patients regarding the patient's autonomy in bathing activities, the material use and the time needed from caregivers in home care. Additionally qualitative data on patient's bathing activities and the use of Showerpatch will be collected.

ELIGIBILITY:
Inclusion Criteria:

* able to read and speak Dutch and to fill out a web-based questionnaire
* patients with an IV catheter (peripheral catheter, midline, peripherally inserted central catheter (PICC), Central Venous catheter (CVC), tunnelled catheter or implantable port) with an expected dwell time IV therapy of at least 14 days and with or without a prospect of discharge to the home setting with the IV catheter in situ in the foreseen study period
* physically able to wash themselves
* with access to the internet

Exclusion Criteria:

* Bedridden patients
* Patients who have already participated in an earlier stage of the ISIC study
* Patients with more than one lumen of the catheter continuously connected to an infusion line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Self-reported autonomy score regarding bathing activities | Weekly until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  autonomy regarding bathing activities will be scored on a newly developed autonomy scale on a weekly basis

SECONDARY OUTCOMES:
Number and type of bathing activities | Weekly reported, until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Number and type of bathing activities per week
Catheter dressing status: wet | Before and after bathing activities, reported until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Expressed on a 3-point scale from 0 which means not wet to 2 totally wet
Catheter dressing status: loose | Before and after bathing activities, reported until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Expressed on a 3-point scale from 0 which means not loose to 2 totally loose
Time needed from a caregiver | Weekly reported, until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Time expressed in minutes per week
Material consumption regarding IV entry site care for bathing activities | Weekly reported, until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Description of material which was used for catheter dressing protection and/or for the extra dressing change and/or extra securement of the dressing afterwards.
Clinical signs of local infection | Before and after bathing activities, reported until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Redness, tenderness, warmth, swelling or pus leakage recorded on a yes/no basis
Laboratory-Confirmed Bloodstream Infection | Until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Collected at the end of the study by retrospective analysis of the patient file in case of hospital admission

OTHER OUTCOMES:
Skin irritation after application of Showerpatch | Before and after bathing activities, reported until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Redness or other sign of skin irritation at the place where adhesive of the new protection dressing had contact with the skin on a yes/no basis
Catheter/Huber needle status | Before and after bathing activities, reported until catheter removal which is expected on an average after 2 weeks or up to 8 weeks
  Expressed on a 3-point scale from 0 which means correct in place to 2 totally removed

CONTACTS AND LOCATIONS:
Overall Officials: Godelieve A Goossens, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Oakley C, Wright E, Ream E. The experiences of patients and nurses with a nurse-led peripherally inserted central venous catheter line service. Eur J Oncol Nurs. 2000 Dec;4(4):207-18. doi: 10.1054/ejon.2000.0099. PMID 12849017
- [Background] Molloy D, Smith LN, Aitchison T. Cytotoxic chemotherapy for incurable colorectal cancer: living with a PICC-line. J Clin Nurs. 2008 Sep;17(18):2398-407. doi: 10.1111/j.1365-2702.2008.02359.x. PMID 18705719
- [Background] Do AN, Ray BJ, Banerjee SN, Illian AF, Barnett BJ, Pham MH, Hendricks KA, Jarvis WR. Bloodstream infection associated with needleless device use and the importance of infection-control practices in the home health care setting. J Infect Dis. 1999 Feb;179(2):442-8. doi: 10.1086/314592. PMID 9878029
- See also: Definition of Laboratory-Confirmed Bloodstream Infection (LCBI) infection — http://www.cdc.gov/nhsn/PDFs/pscManual/4PSC_CLABScurrent.pdf